CLINICAL TRIAL: NCT06229548
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SYH2053 in Subjects With Normal or Elevated Low-Density Lipoprotein Cholesterol
Brief Title: A Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SYH2053
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC Zhongnuo Pharmaceutical (Shijiazhuang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYH2053-001
Record Dates: First submitted 2023-12-20; First posted 2024-01-29 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2023-12

CONDITIONS: Hyperlipemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYH2053 SAD experimental group (Experimental): Subjects in SAD experimental groups will receive a single subcutaneous injection of SYH2053 on Day 1.
  Interventions: Drug: SYH2053
- Placebo SAD group (Placebo Comparator): Subjects in SAD placebo groups will receive a single subcutaneous injection of placebo on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SYH2053 — subcutaneous injection
  Arms: SYH2053 SAD experimental group
Drug: Placebo — subcutaneous injection
  Arms: Placebo SAD group

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single ascending dose (SAD) study of SYH2053 when administered subcutaneously to subjects with normal and elevated LDL-C.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must give informed consent before the trial, fully understand the content, procedures and possible adverse reactions, and voluntarily sign a written informed consent.
2. Sex: male or female subjects.
3. Age of 18 - 60 years (inclusive).
4. BMI: 18.6-28.5 kg/m^2 (inclusive), with a minimum weight of 50 kg (inclusive) for male and 45 kg (inclusive) for female.
5. During screening and baseline, LDL-C ≥100 mg/dL (2.6 mmol/L) and < 190 mg/dL (4.9 mmol/L); TG ≤ 400 mg/dL (4.5 mmol/L); TC < 278 mg/dL (7.2 mmol/L) in serum under fasting state;
6. Subjects have no history of chronic or serious diseases or family history of early-onset coronary heart disease, including cardiovascular, liver, kidney, blood and lymphatic, endocrine, immune, psychiatric, neurological, and gastrointestinal systems, and are generally in good health.
7. The subjects can communicate well with the investigators and complete the trial according to the protocol.

Exclusion Criteria:

1. Allergic constitution or known history of allergy to the components of the study drug or similar drugs.
2. Antibody drugs targeting PCSK9 have been used within 6 months prior to screening, oligonucleotides targeting PCSK9 have been used within 12 months prior to screening.
3. There are currently medical disorders of clinical significance, including but not limited to, circulatory, hematological or hematopoietic diseases, respiratory, endocrine, urinary, digestive, neurological or psychiatric disorders, infections, tumors, severe trauma, or any other diseases that the investigator considers to be excluded or likely to interfere with the interpretation of the findings.
4. Those who underwent major surgery within 6 months prior to initial administration, or who planned to undergo surgery during the study.
5. Clinically significant abnormalities in vital signs, physical examination, electrocardiogram and laboratory examination.
6. The estimated glomerular filtration rate (eGFR) during screening was < 90 mL/min/1.73 m^2 (calculated by simplified MDRD formula).
7. During screening, any item of alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (TBIL), γ-glutamyltransferase (GGT), alkaline phosphatase (ALP) > 1.5×ULN (retest once within 1 week allowed).
8. During screening or baseline, subjects with prolonged QT/QTc interval (QTcF > 450 ms in male, > 470 ms in female).
9. Subjects with non-negative test for any of HBsAg, HCV antibodies, syphilis antibodies, and HIV antibodies.
10. Blood loss or blood donation of more than 200 mL within 3 months prior to administration (except for female menstrual period), and/or platelet donation within 2 weeks prior to administration.
11. Use of any drug, supplement, vitamin or dietary supplement known to affect lipid metabolism within 28 days prior to administration; use of any drug for therapeutic purposes (except topical drugs with local effects) within 14 days prior to administration or within the 7 half-lives of the drug (whichever is longer).
12. A history of drug abuse, and/or drug use within 3 months prior to screening, and/or habitual use of any psychotropic drug, including Chinese herbs.
13. Positive urine drug screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
The Number of Participants with Treatment Related Adverse Events as Assessed by CTCAE v5.0 | Pre-dose and multiple timepoints no less than 57 days
  The investigator will make an assessment of intensity for each AE and SAE reported during the study according to CTCAE V5.0

SECONDARY OUTCOMES:
The serum LDL-C level after dosing SYH2053 | Pre-dose and multiple timepoints no less than 57 days
  measure the LDL-C level in blood by lab examination and evaluate the effect of SYH2053 on LDL-C Level
The serum PCSK9 level after dosing SYH2053 | Pre-dose and multiple timepoints no less than 57 days
  measure the PCSK9 level in blood by lab examination and evaluate the effect of SYH2053 on PCSK9 Level
PK parameters (Cmax) | Pre-dose and multiple timepoints up to 4 days
  maximum peak observed plasma SYH2053 concentration in treated subjects
PK parameters (Tmax) | Pre-dose and multiple timepoints up to 4 days
  time to reach maximum peak plasma SYH2053 concentration in treated subjects
PK parameters (AUC) | Pre-dose and multiple timepoints up to 4 days
  area under the plasma concentration-time curve in SYH2053 treated subjects
PK parameters (T1/2) | Pre-dose and multiple timepoints up to 4 days
  the elimination half-life associated with the terminal slope of a semi-logarithmic concentration-time curve in SYH2053 treated subjects
Immunogenicity of SYH2053 | Pre-dose and multiple timepoints up to 57 days
  Rate of formation of anti-drug antibodies to SYH2053
The serum TC level after dosing SYH2053 | Pre-dose and multiple timepoints no less than 57 days
  measure the TC level in blood by lab examination and evaluate the effect of SYH2053 on TC Level
The serum TG level after dosing SYH2053 | Pre-dose and multiple timepoints no less than 57 days
  measure the TG level in blood by lab examination and evaluate the effect of SYH2053 on TG Level
The serum HDL-C level after dosing SYH2053 | Pre-dose and multiple timepoints no less than 57 days
  measure the HDL-C level in blood by lab examination and evaluate the effect of SYH2053 on HDL-C Level
The serum Lp(a) level after dosing SYH2053 | Pre-dose and multiple timepoints no less than 57 days
  measure the Lp(a) level in blood by lab examination and evaluate the effect of SYH2053 on Lp(a) Level
The serum VLDL-C level after dosing SYH2053 | Pre-dose and multiple timepoints no less than 57 days
  measure the VLDL-C level in blood by lab examination and evaluate the effect of SYH2053 on VLDL-C Level
The serum non-HDL-C level after dosing SYH2053 | Pre-dose and multiple timepoints no less than 57 days
  measure the non-HDL-C level in blood by lab examination and evaluate the effect of SYH2053 on non-HDL-C Level
The serum ApoA1 level after dosing SYH2053 | Pre-dose and multiple timepoints no less than 57 days
  measure the ApoA1 level in blood by lab examination and evaluate the effect of SYH2053 on ApoA1 Level
The serum ApoB level after dosing SYH2053 | Pre-dose and multiple timepoints no less than 57 days
  measure the ApoB level in blood by lab examination and evaluate the effect of SYH2053 on ApoB Level
The serum hsCRP level after dosing SYH2053 | Pre-dose and multiple timepoints no less than 57 days
  measure the hsCRP level in blood by lab examination and evaluate the effect of SYH2053 on hsCRP Level

CONTACTS AND LOCATIONS:
Locations (1):
- 10 Chedaogou Rd.,Haidian District, Beijing, China, Beijing, Beijing Municipality, China